CLINICAL TRIAL: NCT06434324
Title: A Study to Evaluate the Efficacy of Pleural Space Saline Irrigation in Addition to Standard Intrapleural Thrombolytic Therapy in the Management of Empyema/Complicated Parapneumonic Effusion
Brief Title: Pleural Space Saline Irrigation in Addition to Standard Intrapleural Thrombolytic Therapy in Empyema/Complicated Parapneumonic Effusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dagny K. Anderson, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-013234; HT9425-24-C-0010 (Other Grant/Funding Number: US Dept of Defense)
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Pleural Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline Irrigation Group (Experimental): Subjects will receive twice daily fibrinolytic therapy in addition to daily saline irrigation through their chest tube until the treating physician determines that the pleural space has been adequately evacuated
  Interventions: Procedure: Saline Irrigation
- Standard of Care Group (No Intervention): Subjects will receive twice daily fibrinolytic therapy through their chest tube until the treating physician determines that the pleural space has been adequately evacuated

INTERVENTIONS:
Procedure: Saline Irrigation — 250 cc waves of warmed saline irrigation (up to 2000 cc) through thoracostomy tube on a daily basis
  Arms: Saline Irrigation Group

SUMMARY:
The purpose of this study is to see if there is any benefit in adding saline irrigation through a chest tube to the standard course of treatment for people diagnosed or suspected of having a pleural space infection.

DETAILED DESCRIPTION:
Pleural space infections portend considerable morbidity and require procedural and sometimes surgical intervention in the context of prolonged hospital stays (median length of stay has been reported as 14-19 days) for definitive management. Key aspects of management include pleural space evacuation and appropriate antimicrobial therapy. The antimicrobial regimen is initiated intravenously and is often transitioned to an oral regimen as guided by clinical improvement, radiographic improvement, and microbiologic studies though conventional bacterial cultures remain negative in as many as 40% of cases of pleural space infection. There is variability in antimicrobial duration though this is typically continued for at least 3 weeks. The MIST 2 trial investigated the role of intrapleural tissue plasminogen activator (t-PA) and dornase (DNase) in the management of pleural space infections, noting that disrupting septations and reducing pleural fluid viscosity were necessary steps to achieve successful drainage in in-vitro studies. MIST 2 demonstrated that a combination of intrapleural t-PA and DNase improved pleural space evacuation on serial chest x-ray and reduced the frequency of surgical referral and hospital length of stay.

Saline irrigation of the pleural space has been proposed to reduce stasis and dilute bacteria, cytokines, and coagulation factors, which induce pleural space organization. The Pleural Irrigation Trial was a pilot study evaluating the role of 250 cc 0.9% sodium chloride irrigation three times daily for 3 days in comparison to standard care, which included maintaining thoracostomy tubes on suction and flushing with 30 cc three times daily. Saline irrigation led to a 32.3% reduction in pleural fluid volume as assessed by computed tomography in comparison to 15.3% in the standard care arm. Fewer patients in the irrigation group were referred for surgery (OR 7.1).

To our knowledge, the efficacy of intrapleural saline irrigation in addition to fibrinolytic therapy has not been studied in comparison to fibrinolytic therapy alone. The Mayo Clinic Interventional Pulmonary practice in Rochester, MN intends to study this in the context of the inpatient pleural service, the team that is routinely consulted for patients with proven or suspected pleural space infections. This team routinely places and manages ultrasound-guided locking-loop thoracostomy tubes and additionally manages patients with thoracostomy tubes placed by intensivists, surgeons, and interventional radiologists when consulted. Our team intends to recruit hospitalized patients that meet the inclusion/exclusion criteria of the study. Those that provide informed consent to participate in the study will be randomized to usual care versus intrapleural saline irrigation + usual care.

ELIGIBILITY:
Inclusion criteria:

* Purulent pleural fluid versus pleural fluid analysis demonstrating pH <7.2, glucose <60 mg/dL, positive Gram stain, or positive pleural fluid culture versus multiseptated pleural effusion with infection at top of differential diagnosis
* Patients initiating intrapleural lytic therapy under the care of the Interventional Pulmonary consult service at Mayo Clinic in Rochester, MN

Exclusion Criteria:

* Unwillingness to give informed consent
* Patients with known bleeding diathesis
* Platelet count <50,000 per μL
* INR >2.2 (of note, INR can be allowed to drift down or be reversed pharmacologically prior to initiation of intrapleural lytics/saline)
* Current use of systemic anticoagulation or antiplatelet therapy without the ability to hold therapy for the recommended amount of time prior to an invasive procedure (aspirin monotherapy is acceptable)
* Pregnant or nursing females, or females of child-bearing potential who decline a pregnancy test prior to enrollment
* Incarcerated patients
* Presence of ipsilateral bronchopleural fistula
* Current or recent (within past 30 days) presence of tunneled pleural catheter on the same side as the current proven/suspected pleural space infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-29 (Actual); Primary Completion 2026-04-04 (Estimated); Study Completion 2026-05-04 (Estimated)

PRIMARY OUTCOMES:
Adequate pleural space evacuation | Approximately 3 days
  Number of intrapleural fibrinolytic doses to achieve adequate pleural space evacuation (defined as <=2.5 cm separation between parietal and visceral pleural layers on bedside ultrasound or no more than small residual effusion on clinically-directed CT chest imaging).

SECONDARY OUTCOMES:
Need for additional interventions | Approximately 10 days
  Number of additional interventions to achieve satisfactory pleural space evacuation, such as additional paired lytics beyond 6 doses, ipsilateral thoracentesis, additional ipsilateral thoracostomy tube placement, surgical intervention, or discharge with an empyema tube in situ.
Thoracostomy tube days | Approximately 10 days
  Number of thoracostomy tube days from the time that treatment is initiated
Number of hospital days | Approximately 14 days
  Number of hospital days from the time that treatment is initiated
Pain tolerance of pleural space irrigation | Approximately 3 days
  Measured using a visual analog scale (VAS) questionnaire that assesses pain experienced during treatment utilizing a scale of 0 to 10, with 10 meaning the worst pain imaginable.
Number of adverse events | Approximately 10 days
  Total number of adverse events including new/worsened respiratory failure, septic shock, hemothorax

CONTACTS AND LOCATIONS:
Overall Officials: Dagny Anderson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bedawi EO, Ricciardi S, Hassan M, Gooseman MR, Asciak R, Castro-Anon O, Armbruster K, Bonifazi M, Poole S, Harris EK, Elia S, Krenke R, Mariani A, Maskell NA, Polverino E, Porcel JM, Yarmus L, Belcher EP, Opitz I, Rahman NM. ERS/ESTS statement on the management of pleural infection in adults. Eur Respir J. 2023 Feb 2;61(2):2201062. doi: 10.1183/13993003.01062-2022. Print 2023 Feb. PMID 36229045
- [Background] Birkenkamp K, O'Horo JC, Kashyap R, Kloesel B, Lahr BD, Daniels CE, Nichols FC 3rd, Baddour LM. Empyema management: A cohort study evaluating antimicrobial therapy. J Infect. 2016 May;72(5):537-43. doi: 10.1016/j.jinf.2016.02.009. Epub 2016 Mar 15. PMID 26987740
- [Background] Rahman NM, Maskell NA, West A, Teoh R, Arnold A, Mackinlay C, Peckham D, Davies CW, Ali N, Kinnear W, Bentley A, Kahan BC, Wrightson JM, Davies HE, Hooper CE, Lee YC, Hedley EL, Crosthwaite N, Choo L, Helm EJ, Gleeson FV, Nunn AJ, Davies RJ. Intrapleural use of tissue plasminogen activator and DNase in pleural infection. N Engl J Med. 2011 Aug 11;365(6):518-26. doi: 10.1056/NEJMoa1012740. PMID 21830966
- [Background] Mismetti V, Froudarakis ME. Medical management of pleural infection: Why not saline intrapleural lavage? Clin Respir J. 2022 Nov;16(11):693-695. doi: 10.1111/crj.13548. Epub 2022 Sep 29. No abstract available. PMID 36173249
- [Background] Hooper CE, Edey AJ, Wallis A, Clive AO, Morley A, White P, Medford AR, Harvey JE, Darby M, Zahan-Evans N, Maskell NA. Pleural irrigation trial (PIT): a randomised controlled trial of pleural irrigation with normal saline versus standard care in patients with pleural infection. Eur Respir J. 2015 Aug;46(2):456-63. doi: 10.1183/09031936.00147214. Epub 2015 May 28. PMID 26022948
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2024-04-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT06434324/ICF_000.pdf